CLINICAL TRIAL: NCT04320498
Title: Effects of Platelet-rich Plasma in the Treatment of Chronic Anal Fissure
Brief Title: Short Term Results of Platelet-rich Plasma in the Treatment of Chronic Anal Fissure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Yusuf Tanrikulu, Assoc Professor, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122
Record Dates: First submitted 2020-03-12; First posted 2020-03-25 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Anal Fissure Chronic; PRP
Keywords: chronic anal fissure; medical treatment; platelet rich plasma
MeSH Terms: interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): The control patients self-administered topical glyceryl trinitrate, in the perianal area twice a day (Anrecta, Consentis Pharmaceuticals, Istanbul, Turkey)
  Interventions: Drug: Anrecta; Behavioral: sitz bath; Dietary Supplement: nutrition regulation
- PRP group (Experimental): PRP was injected locally in the anal fissure area and glyceryl trinitrate was administered twice daily in the perianal region as in the control group.
  Interventions: Biological: prp injection; Drug: Anrecta; Behavioral: sitz bath; Dietary Supplement: nutrition regulation

INTERVENTIONS:
Biological: prp injection — PRP was injected locally in the anal fissure area and glyceryl trinitrate was administered twice daily in the perianal region as in the control group.
  Other Names: Platelet rich plasma injection
  Arms: PRP group
Drug: Anrecta — self-administered topical glyceryl trinitrate (anrecta), in the perianal area twice a day
  Other Names: rectoderm
Behavioral: sitz bath — participants were told to take a hot water sitz bath once a day
Dietary Supplement: nutrition regulation — The study participants were told to eat a fiber-rich diet and to drink least 2 liters of water daily

SUMMARY:
Autologous PRP currently has many uses in surgical and medical therapy. Compared with other regenerative therapies, PRP is easy-to-prepare, low-cost, and does not require complex equipment. The use of autologous PRP avoids immunological side effects. Data is lacking on the use of PRP in the treatment of anal fissure. This study evaluated PRP as an alternative medical treatment for chronic anal fissures.

DETAILED DESCRIPTION:
. Chronic anal fissures are mucosal ulcers in the anal canal distal to the dentate line and most often present with severe pain and bleeding during defecation. The symptoms of chronic anal fissures persist for more than 8 weeks and do not respond well to medical treatment. This randomized controlled trial investigated the effects of PRP on the healing of chronic anal fissures, which can be considered as nonhealing ulcers. High anal sphincter pressure can cause chronic anal fissures by producing mucosal ischemia in the posterior anal canal that delays wound healing, ultimately resulting in a chronic nonhealing ulcer. Increased anal sphincter pressure induces constipation and spasms in the arterioles that form the mucosal blood supply.9 Botulinum toxin, calcium channel blockers, nitrates, or surgery promote healing by reducing anal sphincter pressure, and increasing blood flow.

Autologous PRP has been shown to speed recovery and improve pain and quality of life scores of patients treated for chronic wounds.PRP reduced complaints and accelerated epithelialization and healing in patients with chronic anal fissures. PRP, which can be obtained easily and did not have any harmful patient effects may be an alternative to surgery in patients with chronic anal fissures. The duration of symptoms should be considered during the evaluation of treatment options.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age with painful defecation of at least 2 months duration and diagnosed with anal fissure between January and October 2019 were included.
* The diagnosis of chronic anal fissure required :
* the presence of internal sphincter muscle fibers in the base of the fissure
* hypertrophic anal papillae on digital rectal examination

Exclusion Criteria:

* Patients with physical examination findings that did not meet the definition of chronic anal fissure
* with painful defecation for less than 2 months,
* atypical fissure location or multiple anal fissures away from the midline
* inflammatory bowel disease
* cancer
* history of trauma
* tuberculosis
* immune suppression
* sexually transmitted disease
* a disease possibly associated with a fissure
* a history of anal surgery
* previous treatment for anal fissure
* current pregnancy .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Between 18 and 65 years of age with chronic anal fissure were included
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
effects of PRP treatment on epithelization . | 10 days , 1 month and 2 months
  In a clean surgical wound, the epithelial cells migrate downward to meet deep in the dermis. Migration ceases when the layer is rejuvenated. Following surgery, this process is normally complete within 48 hours. However, the process of epithelialization is difficult in wounds that are not primarily closed or need to heal by secondary intention. In these wounds, the physical distance of epithelial migration is changed across the length, width, and depth of the wound. In chronic anal fissures, wound epithelization can be evaluated by inspection. Approximately 80 percent of the original strength of the tissue is obtained within six weeks. So we planned to make this assessment on the 10th Day, 1st Month, and 2nd Month for the reason I explained above. We considered the complete epithelization of the fissure as a complete healing. We evaluated patients with epithelialization in the midline but incomplete as partial epithelization.
effect of PRP treatment on VAS scores | 10 days , 1 month and 2 months
  Distribution of the effect of PRP treatment on VAS scores. The VAS is a simple scale with a length of 100 mm on which patients were asked to rate their pain from 0 (absence of pain) to 100 (worst pain imaginable).
  In connection with wound healing, we expect the pain to change. The process of epithelialization is difficult in wounds that are not primarily closed or need to heal by secondary intention. In these wounds, the physical distance of epithelial migration is changed across the length, width, and depth of the wound. So we planned to make this assessment on the 10th Day to evaluate early pain control. we planned In the first month, to evaluate the middle period pain control and in the second month to evaluate the late period pain control.

SECONDARY OUTCOMES:
effect of PRP treatment on symptoms | 10 days , 1 month and 2 months
  Distribution of the effect of PRP treatment on symptoms Presenting symptoms including constipation, pruritus, presence of skin tags, and bleeding was recorded on enrolment. In connection with wound healing, we expect symptoms such as constipation, pruritus, and bleeding to change. we assessed the decline in constipation, pruritus, and bleeding from the start of treatment. we record the symptoms of the patients on the 10th Day, the first month, and the second month. Thus, we compared the response to treatment in the early, middle, and late periods.
Comparison of the effect of treatments on pain according to the onset of symptoms of patients | 10 days , 1 month and 2 months
  The duration of the associated complaints and symptoms distinguishes acute from chronic anal fissures, which are evaluated and treated as conditions with different etiologies and physiology. Acute anal fissures have symptoms of < 8 weeks duration. Chronic anal fissure symptoms have persisted for 8 weeks or longer. The effectiveness of medical treatment changes with time after the appearance of the first anal fissure symptoms and ultimately becomes less effective than surgery. we evaluated the effect of treatments on symptoms according to the onset of symptoms of patients. we evaluated VAS scores on day 10, months 1, and 2 in patients with fissures for less than 12 months than in those with fissures of longer duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Karatay Medicana Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altomare DF, Binda GA, Canuti S, Landolfi V, Trompetto M, Villani RD. The management of patients with primary chronic anal fissure: a position paper. Tech Coloproctol. 2011 Jun;15(2):135-41. doi: 10.1007/s10151-011-0683-7. Epub 2011 May 3. PMID 21538013
- [Background] Gupta PJ. Closed anal sphincter manipulation technique for chronic anal fissure. Rev Gastroenterol Mex. 2008 Jan-Mar;73(1):29-32. PMID 18792671
- [Background] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789
- [Background] Medhi B, Rao RS, Prakash A, Prakash O, Kaman L, Pandhi P. Recent advances in the pharmacotherapy of chronic anal fissure: an update. Asian J Surg. 2008 Jul;31(3):154-63. doi: 10.1016/S1015-9584(08)60078-0. PMID 18658016
- [Background] Wu PI, Diaz R, Borg-Stein J. Platelet-Rich Plasma. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):825-853. doi: 10.1016/j.pmr.2016.06.002. PMID 27788903
- [Background] Dhillon RS, Schwarz EM, Maloney MD. Platelet-rich plasma therapy - future or trend? Arthritis Res Ther. 2012 Aug 8;14(4):219. doi: 10.1186/ar3914. PMID 22894643
- [Background] Li F, Li Q, Wang LF. [Advances in the research of effects of mesenchymal stem cells, exosomes, and platelet-rich plasma in wound repair]. Zhonghua Shao Shang Za Zhi. 2019 Oct 20;35(10):764-768. doi: 10.3760/cma.j.issn.1009-2587.2019.10.012. Chinese. PMID 31658550
- [Background] Etulain J, Mena HA, Meiss RP, Frechtel G, Gutt S, Negrotto S, Schattner M. An optimised protocol for platelet-rich plasma preparation to improve its angiogenic and regenerative properties. Sci Rep. 2018 Jan 24;8(1):1513. doi: 10.1038/s41598-018-19419-6. PMID 29367608
- [Background] Hancock BD. The internal sphincter and anal fissure. Br J Surg. 1977 Feb;64(2):92-5. doi: 10.1002/bjs.1800640204. PMID 890253
- [Background] EISENHAMMER S. The evaluation of the internal anal sphincterotomy operation with special reference to anal fissure. Surg Gynecol Obstet. 1959 Nov;109:583-90. No abstract available. PMID 13819766
- [Background] Notaras MJ. Lateral subcutaneous sphincterotomy for anal fissure--a new technique. Proc R Soc Med. 1969 Jul 7;62(7):713. doi: 10.1177/003591576906200737. No abstract available. PMID 5803521
- [Background] Casillas S, Hull TL, Zutshi M, Trzcinski R, Bast JF, Xu M. Incontinence after a lateral internal sphincterotomy: are we underestimating it? Dis Colon Rectum. 2005 Jun;48(6):1193-9. doi: 10.1007/s10350-004-0914-3. PMID 15906136
- [Background] Kang GS, Kim BS, Choi PS, Kang DW. Evaluation of healing and complications after lateral internal sphincterotomy for chronic anal fissure: marginal suture of incision vs. open left incision: prospective, randomized, controlled study. Dis Colon Rectum. 2008 Mar;51(3):329-33. doi: 10.1007/s10350-007-9122-2. Epub 2008 Jan 4. PMID 18176828
- [Background] Rattan S, Chakder S. Role of nitric oxide as a mediator of internal anal sphincter relaxation. Am J Physiol. 1992 Jan;262(1 Pt 1):G107-12. doi: 10.1152/ajpgi.1992.262.1.G107. PMID 1733256
- [Background] Loder PB, Kamm MA, Nicholls RJ, Phillips RK. 'Reversible chemical sphincterotomy' by local application of glyceryl trinitrate. Br J Surg. 1994 Sep;81(9):1386-9. doi: 10.1002/bjs.1800810949. PMID 7953427
- [Background] Collins EE, Lund JN. A review of chronic anal fissure management. Tech Coloproctol. 2007 Sep;11(3):209-23. doi: 10.1007/s10151-007-0355-9. Epub 2007 Aug 3. PMID 17676270
- [Background] Lund JN, Scholefield JH. A randomised, prospective, double-blind, placebo-controlled trial of glyceryl trinitrate ointment in treatment of anal fissure. Lancet. 1997 Jan 4;349(9044):11-4. doi: 10.1016/S0140-6736(96)06090-4. PMID 8988115
- [Background] Shah V, Lyford G, Gores G, Farrugia G. Nitric oxide in gastrointestinal health and disease. Gastroenterology. 2004 Mar;126(3):903-13. doi: 10.1053/j.gastro.2003.11.046. PMID 14988844
- [Background] Wang HL, Avila G. Platelet rich plasma: myth or reality? Eur J Dent. 2007 Oct;1(4):192-4. No abstract available. PMID 19212466
- [Background] Masoudi E, Ribas J, Kaushik G, Leijten J, Khademhosseini A. Platelet-Rich Blood Derivatives for Stem Cell-Based Tissue Engineering and Regeneration. Curr Stem Cell Rep. 2016 Mar;2(1):33-42. doi: 10.1007/s40778-016-0034-8. Epub 2016 Feb 13. PMID 27047733
- [Background] Schouten WR, Briel JW, Auwerda JJ, De Graaf EJ. Ischaemic nature of anal fissure. Br J Surg. 1996 Jan;83(1):63-5. doi: 10.1002/bjs.1800830120. PMID 8653368
- [Background] Schouten WR, Briel JW, Auwerda JJ. Relationship between anal pressure and anodermal blood flow. The vascular pathogenesis of anal fissures. Dis Colon Rectum. 1994 Jul;37(7):664-9. doi: 10.1007/BF02054409. PMID 8026232
- [Background] Margolis DJ, Kantor J, Santanna J, Strom BL, Berlin JA. Effectiveness of platelet releasate for the treatment of diabetic neuropathic foot ulcers. Diabetes Care. 2001 Mar;24(3):483-8. doi: 10.2337/diacare.24.3.483. PMID 11289472
- [Background] Kazakos K, Lyras DN, Verettas D, Tilkeridis K, Tryfonidis M. The use of autologous PRP gel as an aid in the management of acute trauma wounds. Injury. 2009 Aug;40(8):801-5. doi: 10.1016/j.injury.2008.05.002. Epub 2008 Aug 13. PMID 18703188
- [Background] Dionyssiou D, Demiri E, Foroglou P, Cheva A, Saratzis N, Aivazidis C, Karkavelas G. The effectiveness of intralesional injection of platelet-rich plasma in accelerating the healing of chronic ulcers: an experimental and clinical study. Int Wound J. 2013 Aug;10(4):397-406. doi: 10.1111/j.1742-481X.2012.00996.x. Epub 2012 Jun 4. PMID 22672105
- [Background] Menchisheva Y, Mirzakulova U, Yui R. Use of platelet-rich plasma to facilitate wound healing. Int Wound J. 2019 Apr;16(2):343-353. doi: 10.1111/iwj.13034. Epub 2018 Nov 15. PMID 30440099
- [Background] Motie MR, Hashemi P. Chronic Anal Fissure: A Comparative Study of Medical Treatment Versus Surgical Sphincterotomy. Acta Med Iran. 2016 Jul;54(7):437-40. PMID 27424014
- [Background] Valizadeh N, Jalaly NY, Hassanzadeh M, Kamani F, Dadvar Z, Azizi S, Salehimarzijarani B. Botulinum toxin injection versus lateral internal sphincterotomy for the treatment of chronic anal fissure: randomized prospective controlled trial. Langenbecks Arch Surg. 2012 Oct;397(7):1093-8. doi: 10.1007/s00423-012-0948-2. Epub 2012 Mar 20. PMID 22430300